CLINICAL TRIAL: NCT04550975
Title: Feasibility Randomised Controlled Trial (RCT) of Advanced Cognitive Stimulation Therapy (ACST) for People With Moderate to Severe Dementia
Brief Title: Advanced Cognitive Stimulation Therapy (ACST)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 134729
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: DEM; Dementia; Dementia, Vascular; Dementia, Mixed; Dementia With Lewy Bodies; Dementia Frontal; Dementia Severe; Dementia Moderate; Dementia of Alzheimer Type
Keywords: Dementia; Randomized Controlled Trial; Cognitive Stimulation; Moderate to severe dementia
MeSH Terms: conditions — Dementia; Dementia, Vascular; Mixed Dementias; Lewy Body Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind. Assessor will be blinded to the study. Due to the nature of the intervention, the facilitator and participants cannot be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Cognitive Stimulation Therapy (Experimental): Advanced Cognitive Stimulation Therapy (ACST), a psychosocial intervention, is the modified version of CST for people with moderate and severe dementia. Activities consist of more multisensory stimulation elements than the original CST. ACST will be prescribed to participants 45-minutes per week, biweekly for 7 weeks. The intervention will be delivered by two facilitators, such as a research staff, clinical psychologist trainee or care home staff.
  Interventions: Other: Advanced Cognitive Stimulation Therapy
- Treatment as usual (No Intervention): Standard care in care homes

INTERVENTIONS:
Other: Advanced Cognitive Stimulation Therapy — An adapted version of Cognitive Stimulation Therapy for people with moderate to severe dementia.
  Arms: Advanced Cognitive Stimulation Therapy

SUMMARY:
This study is a feasibility randomised controlled trial (RCT) for an evidence-based intervention for people with moderate to severe dementia. The psychosocial intervention is adapted from Cognitive Stimulation Therapy (CST) and developed within the Medical Research Council (MRC) framework.

DETAILED DESCRIPTION:
The World Health Organization calls for an increase of psychosocial interventions for dementia-a global epidemic. Cognitive Stimulation Therapy (CST) is the only non-pharmacological therapy recommended by the National Institute for Health and Care Excellence for improving cognition for mild to moderate dementia. However, there is little guidance on how to maximise cognition for severe dementia. Advanced Cognitive Stimulation Therapy (ACST) will be the first evidence-based complex intervention for moderate to severe dementia developed within the Medical Research Council (MRC) framework and building upon CST's key principles. This feasibility randomised controlled trial (RCT) aims to 1) evaluate the feasibility of ACST 2) explore if ACST can improve the cognitive function, and QoL, as well as other outcomes including behaviour, engagement, and communication, for people with moderate to severe dementia. A sample of 32 participants will be recruited, where 16 will be randomly allocated to ACST, and 16 to treatment as usual (TAU). Data will be collected pre and post the 7-week intervention period. Improving cognition and QoL for people with moderate to severe dementia is vital because dementia's prevalence is projected to reach 152 million by 2050, resulting in excessive excess disability.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Diagnosis of dementia, according to the DSM-IV
3. SMMSE ≤ 12
4. Ability to communicate in English
5. Ability to complete outcome measures
6. Not having major physical illness or disability that affects participation
7. Consultee is willing and able to provide written informed consent if the participant is not able to provide consent.
8. Ability to remain in a group for around an hour (e.g. no challenging behaviour)

Exclusion Criteria:

1. Illness and disability that affects participation (as deemed by the researcher or attending care home staff)
2. SMMSE < 5
3. Participation in other psychosocial intervention studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment (feasibility of ACST) | Descriptive data will be collected during the study and analysed post-intervention; through study completion, 2 years
  Feasibility of recruitment by successful recruitment of the target sample of 32 in a 24-month period.
Retention rate (feasibility of ACST) | Descriptive data will be collected during the study and analysed post-intervention; through study completion, 2 years
  Retention rate of at least 75% of participants at 8-week follow-up.
Negative or adverse events (acceptability of ACST) | Descriptive data will be collected during the study and analysed post-intervention; through study completion, 2 years
  Any negative or adverse events related to the intervention
Intervention fidelity (acceptability of ACST) | Descriptive data will be collected during the study and analysed post-intervention; through study completion, 2 years
  Facilitator's completion of the fidelity checklist following each session
Intervention fidelity (acceptability of ACST) | Descriptive data will be collected during the study and analysed post-intervention; through study completion, 2 years
  Video recording of all sessions and an independent researcher rating fidelity with a random 10% of the recordings.

SECONDARY OUTCOMES:
Change in cognitive function | Pre test (baseline: week 0) and post test (week 8)
  Exploratory primary outcome; measured pre and post intervention with Standardised Mini-Mental State Examination (Molloy & Standish, 1997) and Test for Severe Impairment (Albert & Cohen, 1992). SMMSE has 11 questions with scores from 0 to 30, where a low score indicates poor performance. TSI has six domains: motor performance, language comprehension, language production, memory, general knowledge, and conceptualisation. Each domain has a maximum score of 4, and a higher score indicates better cognitive ability.
Change in quality of life | Pre test (baseline: week 0) and post test (week 8)
  Exploratory primary outcome; measured pre and post test with Quality of Life in Alzheimer's Disease (QoL-AD) (Logsdon et al., 2002). QoL-AD has 13-items, and a sum score range from 13 to 52; higher score denotes better quality of life.
Change in behaviour | Pre test (baseline: week 0) and post test (week 8)
  Exploratory secondary outcome; measured pre and post test with the Neuropsychiatric Inventory (Cummings et al., 1997). NPI consists of 12 domains. Each question asks for a frequency of symptoms on a 4-point score, severity on a 3-point score, and distress on a 5-point scale. Higher score denotes higher frequency and severity.
Change in communication abilities | Pre test (baseline: week 0) and post test (week 8)
  Exploratory secondary outcome; measured pre and post test with the Holden Communication Scale (Holden & Woods, 1995). Each item contains is on a 5 point scale, and the questionnaire has a maximum score of 48, where a higher score indicates difficulties in communication.
Change in engagement | Evaluated by facilitator after every other session, and independent researcher through recordings; through study completion, up to 24-months
  Exploratory secondary outcome; measured with the Group Observational Measurement of Engagement Tool (Cohen-Mansfield et al., 2017). GOME consists of 5-domains: attendance, engagement, active participation, attitude, and sleep. Each item is measured on a 4- or 7-point Likert scale from 0, none of the time, to 6, all of the time.
Change in overall well-being | Evaluated by assessor through video recordings for every session; through study completion, 2 years
  Exploratory secondary outcome; measured with the Adapted Greater Cincinnati Chapter Well-Being Observation Tool (Adapted GCCWBOT) (Kinney & Rentz, 2005). The facilitator or independent researcher will assess 4 participants at a time. Each evaluation will be 62 minutes, and 8 domains will be assessed: interest, attention, pleasure, self-esteem, normalcy, disengagement, sadness, and negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Spector, PhD, DClinPsych, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: Yes
Study results and IPD will be published in a doctoral thesis, peer-reviewed journals, and presented at conferences, and disseminated to the public through information sheets. Participants who indicate their interest in receiving further information regarding dissemination will be sent a letter with the main findings of the study upon completion. Other researchers can email authors for IPD.
Supporting Information: Study Protocol
Time Frame: Upon study completion
Access Criteria: Email authors

REFERENCES:
- [Background] Molloy DW, Standish TI. A guide to the standardized Mini-Mental State Examination. Int Psychogeriatr. 1997;9 Suppl 1:87-94; discussion 143-50. doi: 10.1017/s1041610297004754. PMID 9447431
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Albert M, Cohen C. The Test for Severe Impairment: an instrument for the assessment of patients with severe cognitive dysfunction. J Am Geriatr Soc. 1992 May;40(5):449-53. doi: 10.1111/j.1532-5415.1992.tb02009.x. PMID 1634695
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Wood S, Cummings JL, Hsu MA, Barclay T, Wheatley MV, Yarema KT, Schnelle JF. The use of the neuropsychiatric inventory in nursing home residents. Characterization and measurement. Am J Geriatr Psychiatry. 2000 Winter;8(1):75-83. doi: 10.1097/00019442-200002000-00010. PMID 10648298
- [Background] Cohen-Mansfield J, Hai T, Comishen M. Group engagement in persons with dementia: The concept and its measurement. Psychiatry Res. 2017 May;251:237-243. doi: 10.1016/j.psychres.2017.02.013. Epub 2017 Feb 6. PMID 28214783
- [Background] Kinney JM, Rentz CA. Observed well-being among individuals with dementia: Memories in the Making, an art program, versus other structured activity. Am J Alzheimers Dis Other Demen. 2005 Jul-Aug;20(4):220-7. doi: 10.1177/153331750502000406. PMID 16136845
- [Background] Holden UP, Woods RT. Positive approaches to dementia care. Edinburgh: Churchill Livingstone, 1995.